CLINICAL TRIAL: NCT01773720
Title: Evaluation of Reliability of Cardiac Output Monitoring Based on Uncalibrated Pulse Contour Analysis During Off-pump Coronary Artery Bypass Grafting
Brief Title: Reliability of Cardiac Output Monitoring Based on Uncalibrated Pulse Contour Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northern State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: UncalPCA-vs-TPTD
Record Dates: First submitted 2013-01-15; First posted 2013-01-23 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Cardiac Index
Keywords: cardiac index; coronary artery bypass; uncalibrated pulse contour analysis; hemodynamic monitoring

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — No biospecimens are to be retained.
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of our study was to evaluate the reliability of uncalibrated cardiac index monitoring based on arterial waveform analysis in patients undergoing off-pump coronary artery bypass grafting.

DETAILED DESCRIPTION:
Using contemporary statistical method the cardiac index values obtained via uncalibrated pulse contour analysis with Pro AQT system will be compared with traditional transpulmonary thermodilution technique (Pulsion, Germany).

ELIGIBILITY:
Inclusion Criteria:

* elective off-pump coronary artery bypass grafting

Exclusion Criteria:

* age < 18 and > 80 years,
* preoperative ejection fraction < 0.35,
* severe cardiac valve dysfunction or peripheral vascular disease,
* constant atrial fibrillation,
* simultaneous interventions (carotid endarterectomy, aneurysm repair, etc.),
* transfer to cardiopulmonary bypass.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease, ranked ASA II-III and scheduled for elective off-pump coronary artery bypass grafting
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Validity of cardiac index measurement | Up to 24 hrs post surgery
  Accuracy and precision of cardiac index measurement using uncalibrated pulse contour analysis in comparison with transpulmonary thermodilution

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Y Kirov, MD, PhD, Study Director — Northern State Medical Univercity
Locations (1):
- Dep. of Anesthesiology, Northern SMU, Arkhangelsk, Russia

REFERENCES:
- [Derived] Smetkin AA, Hussain A, Kuzkov VV, Bjertnaes LJ, Kirov MY. Validation of cardiac output monitoring based on uncalibrated pulse contour analysis vs transpulmonary thermodilution during off-pump coronary artery bypass grafting. Br J Anaesth. 2014 Jun;112(6):1024-31. doi: 10.1093/bja/aet489. Epub 2014 Feb 13. PMID 24531685